CLINICAL TRIAL: NCT00432770
Title: A Phase 1, Single-Site, Double-Blind,Randomized, Dose Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Intravenous Bolus or Intravenous Bolus Followed by Continuous Infusion Administration of ARC1779 Compared to Placebo in Healthy Volunteers
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics of ARC1779 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Archemix Corp. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1779-06-001
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — ARC 1779

INTERVENTIONS:
Drug: ARC1779

SUMMARY:
The purpose of this study is to establish the overall safety and tolerability of ARC1779 in healthy volunteers, and to characterize its pharmacokinetic and pharmacodynamic profile with respect to parameters of platelet function and von Willebrand Factor activity.

DETAILED DESCRIPTION:
The purpose of this study is to establish the overall safety and tolerability of ARC1779 in healthy volunteers, and to characterize its pharmacokinetic and pharmacodynamic profile with respect to parameters of platelet function and von Willebrand Factor activity.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 to ≤ 65 years of age
* Weight ≤ 110 kg
* Negative qualitative urine drug/alcohol test
* Female volunteers must be of non-childbearing potential
* Male volunteers must agree to use a medically acceptable contraceptive
* Volunteers must be capable of understanding and complying with the protocol and must have signed the informed consent document

Exclusion Criteria:

Any clinically significant medical disorder (e.g. diabetes, hypertension, etc.)

* Tendency to bleed easily
* History of recent trauma or surgery
* History of gout or renal stones

Clinically significant abnormal lab parameters for the following:

* PT INR > 1.4
* aPTT > reference laboratory values
* Serum creatinine > 1.3 mg/dL
* Platelet count of ≤ 100,000/mm3
* ALT/AST > 2 times ULN
* WBC ≤ 3000 x 109/L
* Hemoglobin < 11 g/dL
* Total bilirubin > 1.2 mg/dL
* CBT > 15 min

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2006-12; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bioanalytical Systems, Inc, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581
- [Derived] Gilbert JC, DeFeo-Fraulini T, Hutabarat RM, Horvath CJ, Merlino PG, Marsh HN, Healy JM, Boufakhreddine S, Holohan TV, Schaub RG. First-in-human evaluation of anti von Willebrand factor therapeutic aptamer ARC1779 in healthy volunteers. Circulation. 2007 Dec 4;116(23):2678-86. doi: 10.1161/CIRCULATIONAHA.107.724864. Epub 2007 Nov 19. PMID 18025536